CLINICAL TRIAL: NCT02414230
Title: F 18 T807 Tau PET Imaging in Familial Amyotrophic Lateral Sclerosis (IND 123119 Protocol B)
Brief Title: F 18 T807 Tau PET Imaging in Familial Amyotrophic Lateral Sclerosis
Acronym: T807ALS
Status: Completed | Type: Observational
Sponsor: Tammie L. S. Benzinger, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Tammie L. S. Benzinger, MD, PhD, Professor of Radiology and Neurological Surgery, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Other Study IDs: IND 123119 Protocol B
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: fronto-temporal dementia; Tauopathies; Nervous System Diseases; Neurodegenerative Diseases
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Tauopathies; Nervous System Diseases; Neurodegenerative Diseases | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Experimental F 18 T807
  Interventions: Drug: Drug: F 18 T807

INTERVENTIONS:
Drug: Drug: F 18 T807 — Participants will receive a single intravenous bolus injection of approximately 6.5-10mCi (240-370MBq) of F 18 T807. For those who cannot tolerate the full exam, participants will receive single intravenous bolus injection of approximately 6.5-10mCi (240-370MBq) of F 18 T807.
  Other Names: Drug: 18F-AV-1451

SUMMARY:
The purpose of this research study is to evaluate tau distribution in the brain of subjects with: ALS caused by different genetic mutations, any mutation carriers (with or without symptoms), any non-mutation carrier, any sporadic FTD, normal controls.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants, at least 18 years of age.
2. Clinically diagnosed with amyotrophic lateral sclerosis (ALS), fronto-temporal dementia (FTD), or both; or a carrier of a mutation known to cause ALS or FTD (with or without symptoms); or a normal control.
3. Participant is able and willing to undergo testing (psychometric testing, MRI or CT, PET, radioactive tracer injection; for those unable to undergo an MRI, CT will be used to generate regions-of-interest).
4. Pre-menopausal women will undergo a urine pregnancy test within 24 hours of drug administration.

Exclusion Criteria:

1. Has any condition that, in the Investigator's opinion, could increase risk to the participant, limit the participant's ability to tolerate the experimental procedures, or interfere with the collection/analysis of the data (for example, participants with significant respiratory involvement may not be able to lie flat during the scanning procedures).
2. Is deemed likely unable to perform the imaging procedures for any reason.
3. Has a high risk for Torsades de Pointes or is taking medications known to prolong QT interval.
4. Has hypersensitivity to F 18 T807 or any of its excipients.
5. Contraindications to PET, PET-CT or MR (e.g. electronic medical devices, inability to lie still for long periods) that make it unsafe for the individual to participate.
6. Severe claustrophobia.
7. Currently pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Collaborating neuromuscular physicians will refer participants for MR and PET imaging to evaluate tau distribution in the brain of subjects with ALS, or ALS with frontotemporal dementia caused by different genetic mutations, or any mutation carrier (with or without symptoms), or normal controls.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-09-19 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
F 18 T807 Standard Uptake Value Ratios (SUVR) will be correlated with other imaging modalities (MRI, PET amyloid imaging) and cognitive performance. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tammie Benzinger, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share the data with other researchers. They may be doing research in areas similar to this research or in other unrelated areas. These researchers may be at Washington University, at other research centers and institutions, or industry sponsors of research. We may also share this research data with large data repositories (a repository is a database of information) for broad sharing with the research community. If the individual research data is placed in one of these repositories only qualified researchers, who have received prior approval from individuals that monitor the use of the data, will be able to look at the information.

REFERENCES:
- [Result] Ly CV, Koenig L, Christensen J, Gordon B, Beaumont H, Dahiya S, Chen J, Su Y, Nelson B, Jockel-Balsarotti J, Drain C, Jerome G, Morris JC, Fagan AM, Harms MB, Benzinger TLS, Miller TM, Ances BM. Tau positron emission tomography imaging in C9orf72 repeat expansion carriers. Eur J Neurol. 2019 Sep;26(9):1235-1239. doi: 10.1111/ene.13940. Epub 2019 Mar 25. PMID 30790403

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT02414230/Prot_SAP_000.pdf